CLINICAL TRIAL: NCT00002985
Title: Double-Blind Randomized Evaluation of Clinical Benefits of DOXIL in Patients With AIDS-Related Kaposi's Sarcoma Treated With DOXIL or DaunoXome
Brief Title: Doxorubicin in Treating Patients With AIDS-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: DS 96-28; RPCI-DS-96-28; SEQUUS-30-38; NCI-G97-1241
Record Dates: First submitted 1999-11-01; First posted 2004-05-19 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: Sarcoma
Keywords: AIDS-related Kaposi sarcoma
MeSH Terms: conditions — Sarcoma; AIDS-related Kaposi sarcoma | interventions — Daunorubicin

INTERVENTIONS:
Drug: daunorubicin hydrochloride
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether doxorubicin is more effective than daunorubicin for AIDS-related Kaposi's sarcoma.

PURPOSE: Randomized double-blinded phase III trial to determine if doxorubicin is more effective than daunorubicin in treating patients who have AIDS-related Kaposi's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the clinical benefit of doxorubicin HCl liposome (Doxil) compared to baseline status in the treatment of AIDS-related Kaposi's sarcoma. II. Determine tumor response to Doxil as a corollary to clinical benefit. III. Evaluate the safety of Doxil.

OUTLINE: This is a randomized, prospective, double blind, multicenter study. Patients are randomly assigned to receive doxorubicin HCl liposome (Doxil) or daunorubicin (DaunoXome) in a 3:1 ratio. Both Doxil and DauonoXome are given every 2 weeks for 6 courses by intravenous infusion over 60 minutes into a peripheral vein.

PROJECTED ACCRUAL: 80 patients will be studied.

ELIGIBILITY:
DISEASE CHARACTERISTICS: AIDS-related Kaposi's sarcoma that requires systemic chemotherapy One or more of the following (Kaposi's sarcoma- or AIDS-associated): Edema that impairs functional activity Symptomatic, evaluable pulmonary Kaposi's sarcoma documented within 3 months before study Symptomatic, evaluable GI Kaposi's sarcoma documented within 3 months before study Moderate or severe pain despite the use of analgesics Lesion(s) that patient feels are disfiguring and impair patient's self-image or daily activities At least 5 bidimensionally measurable monocutaneous lesions

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Karnofsky 40-100% Life expectancy: At least 120 days Hematopoietic: Neutrophil count at least 1,200 cells/mm3 Platelet count at least 75,000 cells/mm3 Hemoglobin at least 9.0 g/dL Hepatic: Creatinine less than 2 times upper limit of normal (ULN) Bilirubin less than 2 times ULN Renal: Not specified Cardiovascular: Cardiac ejection fraction at least 50% No histopathological evidence of antracycline-induced cardiomyopathy Pulmonary: No significant non-Kaposi's sarcoma associated pulmonary insufficiency (defined as oxygen saturation less than 90%) Other: Not pregnant or nursing Fertile women must be using medically proven method of birth control No opportunistic infection in the past 4 weeks No other active malignancies except basal or squamous cell carcinoma of the skin or in situ cervical or anal carcinoma No neuropsychiatric history or altered mental status that prevents informed consent or compliance with protocol requirements

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 14 days since prior anti-Kaposi's sarcoma therapy No prior Doxil or DaunoXome No concurrent cytotoxic chemotherapy Endocrine therapy: Not specified Radiotherapy: No concurrent radiation therapy Surgery: Not specified Other: Antiviral therapy allowed Colony stimulating factors allowed Erythropoietin allowed Prophylactic therapy, maintenance therapy and treatment for HIV-associated opportunistic infections allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-11; Primary Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence P. Leichman, MD, Study Chair — Albany Medical College
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States